CLINICAL TRIAL: NCT05354648
Title: Effects of Hypoxic-hyperoxic Preconditioning on Myocardial Protection Against Ischemia-reperfusion Injury in Cardio-surgical Patients
Brief Title: Effects of Hypoxic-hyperoxic Preconditioning in Cardio-surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Research Clinical Center of Federal Medical & Biological Agency, Russia (Other Government)
Collaborators: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other); Siberian State Medical University (Other); I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HHP-cardio
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: Myocardial Reperfusion Injury; Hypoxia; Hyperoxia; Coronary Artery Disease
Keywords: myocardial protection; preconditioning; hypoxia; hyperoxia; ischemia-reperfusion injury; cardiopulmonary bypass; oxygen transport
MeSH Terms: conditions — Myocardial Reperfusion Injury; Hypoxia; Hyperoxia; Coronary Artery Disease; Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypoxic-hyperoxic preconditioning (HHP) (Active Comparator): HHP was carried out as follows: breathing with a hypoxic gas mixture for 10 min with the development of hypoxemia, then breathing with a hyperoxic gas mixture for 30 minutes, and at the last stage, a period of breathing with atmospheric air until the cardio-pulmonary bypass is connected. The anaerobic threshold was determined 72 hours before surgery to establish a safe oxygen concentration in the respiratory gas mixture during the hypoxic phase of preconditioning.
  Interventions: Procedure: Hypoxic-hyperoxic preconditioning
- Control (Placebo Comparator): The anaerobic threshold was determined, however, patients in the control group were not preconditioned. Mechanical ventilation was carried out with individual settings maintaining the target values of PaO2 and PaCO2 (80 - 120 mm Hg and 35 - 45 mm Hg, respectively), until the cardio-pulmonary bypass was connected.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Hypoxic-hyperoxic preconditioning — Patients were intubated and mechanically ventilated with the target values of PaO2 and PaCO2 (80 - 120 mm Hg and 35 - 45 mm Hg, respectively) under the inhalation anesthesia. HHP was carried out as follows: breathing with a hypoxic gas mixture for 10 min with the development of hypoxemia, then breathing with a hyperoxic gas mixture for 30 minutes, then a period of breathing with atmospheric air (normoxia and normocapnia) until the cardio-pulmonary bypass is connected.
  Other Names: HHP
  Arms: Hypoxic-hyperoxic preconditioning (HHP)
Procedure: Placebo — Patients were intubated and mechanically ventilated with the target values of PaO2 and PaCO2 (80 - 120 mm Hg and 35 - 45 mm Hg, respectively) under the inhalation anesthesia until the cardio-pulmonary bypass is connected.
  Arms: Control

SUMMARY:
Coronary artery bypass grafting (CABG) with cardiopulmonary bypass is a common surgical therapy for patients suffering from coronary artery diseases. The heart is subjected to a long period of ischemia due to the occlusion of the aorta. The heavy burden of myocardial ischemia-reperfusion injury (IRI) thus induces cardiomyocyte death, which can paradoxically reduce the beneficial effect of CABG. Preconditioning by moderate hypoxia or hyperoxia serves as an effective drug-free method to increase the organism's resistance to negative effects, including IRI.

DETAILED DESCRIPTION:
It has been firmly established that the diminished oxygen delivery to the tissues in response to hypoxia is countered by a combination of the increased regional blood flow and the enhanced functional capillary density in the microcirculation. In experimental studies, exposure to hyperoxia for a limited time before ischemia induces a low-grade systemic oxidative stress evokes a preconditioning-like effect on the myocardium and reduces the infarction area by 20%, and the number of arrhythmias after ischemia-reperfusion. One hundred twenty patients were randomly assigned into two equal groups: hypoxic-hyperoxic preconditioning before the surgery (HHP group) and the control group (without preconditioning). Safety control of the preconditioning procedure included ECG monitoring, invasive blood pressure, cardiac output, pulse oximetry, capnography, cerebral oximetry, measurement of anaerobic threshold; acid-base status and metabolic state of arterial and venous blood were assessed once every 10 min during the preconditioning procedure; oxygen balance parameters were calculated. Seventy-two hours before the surgery, an anaerobic threshold was determined to establish a safe oxygen concentration in the respiratory gas mixture during the hypoxic preconditioning phase from 10 to 14%, followed by 75-80% oxygen concentration during the hyperoxic phase.

The hypoxic-hyperoxic preconditioning with individual parameters selection based on the anaerobic threshold in patients with coronary artery diseases before the main stage of cardiac surgery with a cardiopulmonary bypass should reduce the duration of mechanical ventilation, catecholamine support, and frequency of perioperative complications.

ELIGIBILITY:
Inclusion Criteria:

* the need for coronary artery bypass grafting (CABG)

Exclusion Criteria:

* age over 75 years
* emergency surgery
* diabetes mellitus
* exacerbation of a chronic disease 1 week before surgery
* any oncological disease at the time of the examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-01-15 (Actual); Study Completion 2016-02-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants with complications | 60 days
  Any type of complications in postoperative period
Mechanical ventilation | 60 days
  Mechanical ventilation time
Rate of spontaneous sinus rhythm recovery | 14 days
  Spontaneous sinus rhythm recovery after surgery

SECONDARY OUTCOMES:
Catecholamine support | 60 days
  Catecholamine support time
Troponin T | 12 hours
  Troponin T concentration
Endothelin-1 | 1 day before surgery
  Endothelin-1 concentrations
Endothelin-1 dynamics 1 | at the end of surgery
  Endothelin-1 concentrations
Endothelin-1 dynamics 2 | 24 hours after surgery
  Endothelin-1 concentrations
NOx total | 1 day before surgery
  NOx total concentrations
NOx total dynamics 1 | at the end of surgery
  NOx total concentrations
NOx total dynamics 2 | 24 hours after surgery
  NOx total concentrations
Asymmetric dimethylarginine (ADMA) | 1 day before surgery
  ADMA concentrations
ADMA dymanics 1 | at the end of surgery
  ADMA concentrations
ADMA dymanics 2 | 24 hours after surgery
  ADMA concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Irina A Mandel, PhD, Principal Investigator — Federal Research Clinical Center FMBA Russia

REFERENCES:
- [Background] Mandel IA, Podoksenov YK, Suhodolo IV, An DA, Mikheev SL, Podoksenov AY, Svirko YS, Gusakova AM, Shipulin VM, Yavorovskiy AG. Influence of Hypoxic and Hyperoxic Preconditioning on Endothelial Function in a Model of Myocardial Ischemia-Reperfusion Injury with Cardiopulmonary Bypass (Experimental Study). Int J Mol Sci. 2020 Jul 27;21(15):5336. doi: 10.3390/ijms21155336. PMID 32727110